CLINICAL TRIAL: NCT05350202
Title: Empagliflozin Functional Capacity - Non-Interventional Study
Brief Title: Emp-Activity: Empagliflozin Functional Capacity
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0259
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Empagliflozin-treated patients: Patients with heart failure (HF), with or without diabetes, who received their first prescription of empagliflozin were treated according to the approved product information, with a recommended daily dose of 10 milligrams (mg).
  Interventions: Drug: Empagliflozin
- Non-SGLT2i-treated patients: Patients with heart failure (HF), with or without diabetes, who received drugs with mechanisms of action other than empagliflozin (drugs other than SGLT2i (Sodium-Glucose Co-Transporter 2 inhibitors)) were treated according to the approved product information.

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin was administered according to the approved product information.
  Other Names: Jardiance®
  Groups: Empagliflozin-treated patients

SUMMARY:
This is a multinational non-interventional study based on newly collected data to assess demographics, disease, and treatment pattern of patients with chronic Heart Failure (HF) in a two-cohort design: one cohort will receive first prescription of empagliflozin as routine therapy for HF, the other cohort will receive HF therapy with drugs with another mechanism of action. Treatment of HF according to routine practice is determined by the physician independent of the participation of the patient in this non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to study participation
* Male and female patients ≥ 18 years at Visit 1
* Patients must be contractually capable and mentally able to understand and follow the instructions of the study personnel
* Patients with diagnosis of chronic heart failure NYHA Class 2-4
* Treatment-naïve for SGLT2i at visit 1
* Women of childbearing potential must take appropriate precautions against getting pregnant according to approval of chosen HF drug(s)

Exclusion Criteria:

* Missing physician's diagnosis of chronic heart failure
* Patients hospitalized at visit 1
* Life expectancy ≤ 12 months according to physician's assessment
* Lack of informed consent
* Pregnant or lactating females
* Participation in a parallel interventional clinical trial
* Chosen treatment with another SGLT2i drug than empagliflozin
* Having been enrolled into the non-empagliflozin-arm of this non-interventional study
* Current or prior treatment with SGLT2i at visit 1
* Patients with contraindications according to current Summary of Product Characteristics (SmPC)
* Patients with dependency or relationship to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic Heart Failure (HF) in a two cohort design: one cohort will receive first prescription of empagliflozin as routine therapy for HF, the other cohort will receive HF therapy with drugs with another mechanism of action.
Sampling Method: Non-Probability Sample
Enrollment: 3431 (Actual)
Dates: Start 2022-12-18 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (349):
- Bulgaria (35):
  - Dr. Mircheva, Burgas
  - Dr. Yordanov, Haskovo
  - MBAL Atanas Dafovski, Kardzhali, Kardzhali
  - Dr. Krasteva, Kyustendil
  - Dr. Todorov, Lovech
  - Dr. Tsoneva, Lovech
  - Dr. Pavlov, Parvomay
  - Medical Center, Pazardjik, Pazardzhik
  - Dr. Stankova, Pernik
  - assoc.prof. Gospodinov, Pleven
  - dr. Kostadinovska, Pleven
  - prof.Tisheva, Pleven
  - Dr. Mekenian, Plovdiv
  - Dr. Ilchev, Plovdiv
  - Dr. Hairabedian, Plovdiv
  - Dr. Filipov, Plovdiv
  - MBAL Sliven, Dr. Bletsova, Sliven
  - Dr. Pancheva, Sofia
  - prof. Velchev, Sofia
  - dr. Georgieva, Sofia
  - dr. Karchinova, Sofia
  - prof.Vitlianova, Sofia
  - dr. Petrusheva, Sofia
  - dr. Garvanski, Sofia
  - Dr. Naidenova, Sofia
  - Dr. Varnaliiska, Sofia
  - prof. Karamfiloff, Sofia
  - Dr. Nossikov, Sofia
  - Dr. Gospodinov, Stara Zagora
  - Dr. Trendafilova, Targovishte
  - dr. Belcheva, Varna
  - dr. Mancheva, Varna
  - dr. Gyuzelev, Varna
  - Dr. Petrova, Yambol
  - Dr. Toneva-Zhelaeva, Yambol
- Czechia (41):
  - MUDr. Hana Burianová, Bílovec
  - Fakultní nemocnice u sv. Anny v Brně, Brno
  - MUDr. Karel Kameník s.r.o., Brno
  - MUDr. Libor Nechvátal s.r.o., Brno
  - Zdravá srdce s.r.o., Brno
  - Kardiologická ambulance Brno, s.r.o., Brno-Královo Pole
  - EDUMED s.r.o. - Dr. Nováková, Broumov
  - EDUMED s.r.o. - Dr. Polášková, Broumov
  - EDUMED s.r.o. - Dr. Švarcová, Broumov
  - EDUMED s.r.o., Broumov
  - Kardiologická ambulance Český krumlov, Český Krumlov
  - CorMedico s.r.o., Frýdek-Místek
  - DIKa centrum s.r.o., Havířov
  - Lékařský servis, a.s., Havířov
  - Kardio Pudich s.r.o., Hlučín
  - ProKardio HK, s.r.o., Hradec Králové
  - Nemocnice Jihlava - Kardiologické oddělení, Jihlava
  - Oblastní nemocnice Kolín, a.s. nemocnice Středočeského kraje, Kolín
  - KardioBušák s.r.o., Louny
  - Kardiomost s.r.o., Most
  - Nemocnice AGEL Nový Jičín, a.s., Nový Jičín
  - Kardiologická ambulance Olomouc, Olomouc
  - Nemocnice AGEL Ostrava-Vítkovice a.s. - Kardiologická ambulance, Ostrava
  - Kardiologická ambulance Mammed, Ostrava
  - OVAKARD s.r.o., Ostrava
  - Poliklinika Nová Huť, Ostrava
  - Fakultní nemocnice Ostrava, Ostrava - Poruba
  - Kardiologie Vinohrady s.r.o., Prague
  - Kardiologie prof. Táborský s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - MEDICON a.s., Prague
  - Nemocnice na Homolce, Prague
  - Clinical Trials Service s.r.o., Prague
  - ROcardia s.r.o., Prostějov
  - Galenica Medical s.r.o., Prostřední Suchá
  - KARDIO GRÉZL, s.r.o., Šumperk
  - Všeobecná interní ambulance s.r.o., Tábor
  - Kardiologická ambulance MUDr. Ferkl s.r.o., Trutnov
  - Nemocnice AGEL Třinec-Podlesí a.s., Třinec Podlesí
  - Lunacor s.r.o., Vizovice
  - Krajská nemocnice T. Bati, a.s., Zlín
- Hungary (13):
  - Állami Szívkórház, Balatonfüred
  - Gottsegen György National Cardiovascular Center, Budapest
  - Heart and Vascular Centre, Semmelweis University, Budapest
  - Sante Cons Bt., Budapest
  - DE Klinikai Központ Kardiológia és Szívsebészet, Debrecen
  - Dombóvári Szent Lukács Kórház, Dombóvár
  - Lahynara Bt, Dunavarsány
  - Kardiológia Magánrendelő, Eger
  - Mohácsi Kórház, Mohács
  - Coromed-Smo, Pécs
  - University of Pécs, Pécs
  - Soproni Erzsébet Oktató Kórház, Sopron
  - Újszeged Egészségközpont, Szeged
- Poland (115):
  - ECHOKardio Poradnia Kardiologiczna, Bialystok
  - Klinika Kardiologii Uniwersyteckiego Szpitala Klinicznego w Białymstoku, Bialystok
  - Kardiologiczna Praktyka Lekarska Anna Tomaszuk-Kazberuk, Bialystok
  - Podlaski Ośrodek Kardiologii, Bialystok
  - Specjalistyczna Praktyka Lekarska Marek Styczkiewicz, Brzozów
  - BlueMed - Centrum Medyczne, Bydgoszcz
  - Centrum Kardiologii Paweł Grzelakowski, Bydgoszcz
  - Centrum Medyczne A i D Nowak sj, Bydgoszcz
  - Indywidualna Specjalistyczna Praktyka Lekarska Tomasz Ługowski, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska Grzegorz Grześk, Bydgoszcz
  - Indywidualna Specjalistyczna Praktyka Lekarska Jolanta Nowak, Bytom
  - Specjalistyczna Praktyka Lekarska Agata Fenger, Chorozow
  - Med. - Zone sp zoo, Cieszyn
  - Specjalistyczna Praktyka Lekarska lek.n.med.Lucyna Góras-Hetmańczyk, Czeladź
  - Gabinet Kardiologiczny - Jacek Jafra, Częstochowa
  - Prywatna Praktyka Lekarska Artur Dekiela, Częstochowa
  - Specjalistyczna Praktyka Lekarska Magdalena Miczko, Dąbrowa Górnicza
  - ISPL Małgorzata Dobrowolska Gabinet Tendo, Gdynia
  - Specjalistyczna Praktyka Lekarska Wojciech Czapla, Gliwice
  - Dorota Adamczyk-Kot NZOZ-KARDIO, Gmina Jędrzejów
  - Lekarze na Dworskiej, Gmina Świebodzin
  - Indywidualna Praktyka Lekarska Tomasz Zieliński, Grodzisk Mazowiecki
  - Przychodnia Lekarska Zdrowy Miś, Grójec
  - Miedziowe Centrum Zdrowia S.A., Głogów
  - Centrum Medyczne NIWA, Głogów Małopolski
  - Indywidualna Praktyka Lekarska Piotr Tokarczyk, Inowrocław
  - Familia Medicina Sp. z o.o., Iwanowice Włościańskie
  - Specjalistyczna Praktyka Lekarska Urszula Winiarska-Waluś, Jastrzębie Zdrój
  - Specjalistyczna Praktyka Lekarska Jarosław Paździerz, Jasło
  - Centrum Medyczne Kinesis, Kamień
  - Praktyka Lekarska Wojciech Kwaśniewski, Katowice
  - Prywatna Przychodnia Specjalistyczna Drozd Zbigniew Gąsior, Katowice
  - CUM PromontMed, Kielce
  - Arsmedica Specjalistyczna Praktyka Lekarska lek.med. Krzysztof Czerniejewski, Konin
  - Prywatny Gabinet Kardiologiczny lek. med. Sławomir Kępski, Konin
  - Specjalistyczna Praktyka Lekarska Paweł Michalski, Konin
  - Uromed Sp Zoo, Koszalin
  - Poliklinika MSWiA/Indywidualna Specjalistyczna Praktyka Lekarska Krzysztof Jarząbek, Koszalin
  - Indywidualna Praktyka Lekarska Krzysztof Maślak, Koźminek
  - Centrum Medyczne Dietla 19 sp. Z o.o., Krakow
  - Centrum Twojego Zdrowia, Krakow
  - Specjalistyczna Praktyka Lekarska "Kardiolek" Dr med. Piotr Wilkołek, Krakow
  - CM Oficerskie, Krakow
  - Poradnia Kardiologiczna, Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Prywatny Gabinet Kardiologiczny Dr n.med Janusz Bąk, Kranse
  - Centrum Medyczne Dębina, Krościenko Wyżne
  - Beata Mikłaszewicz&Dariusz Dąbrowski Cardiamed S.J., Legnica
  - NZOZ DUOMED S.C. Poradnia Kardiologiczna, Legnica
  - Prywatny Specjalistyczny Gabinet Kardiologiczno-Internistyczny, Libiąż
  - Santa Sp. z o.o., Lodz
  - Nzoz Salusmed, Lodz
  - Kardiologiczna Praktyka Lekarska Wojciech Kula, Lublin
  - NZOZ Sanus Jacek Madej Poradnia kardiologiczna, Lublin
  - NZOZ Sanus Jacek Madej, Lublin
  - Provivo Specjalistyczne Centrum Medyczne, Lublin
  - Indywidualna Specjalistyczna Praktyka Lekarska - Renata Leniec, Lublin
  - Niepubliczny Zakład Opieki Zdrowotnej Specjalistyczne Gabinety lekarskie, Mikołów
  - Gabinet Lekarski Kardiologiczny, Mirków
  - Prywatne Usługi Medyczne Jacek Morka, Modliszewice
  - Indywidualna Specjalistyczna PraktyKa Lekarska-Piotr Utz, Moszczenica
  - Gabinet Lekarski Ewa Burchard, Nowe Miasto nad Pilicą
  - Medyczne Centrum Zdrovita, Nowy Tomyśl
  - Oleśnica Prywatna Praktyka Lekarska, Oleśnica
  - SZOZ Jantar Sp. z o.o. Poradnia Lekarzy Specjalistów, Ostrów Wielkopolski
  - GVM CARINT Oświęcim, Oświęcim
  - Specjalistyczna Praktyka Lekarska Rafał Nowak, Piasek
  - Specjalistyczna Praktyka Lekarska Andrzej Bęben, Piotrkow Trybunalski
  - Indywidualna Specjalistyczna Praktyka Lekarska Andrzej Bolewski, Poznan
  - Wojewódzki Szpital im. św. Ojca Pio w Przemyślu, Przemyśl
  - Leszek Kaminski Specjalistyczny Gabinet Lekarski, Przeworsk
  - Praktyka Lekarska Katarzyna Czarnecka, Pszczyna
  - PCK - Puławskie Centrum Kardiologiczne Przychodnia Specjalistyczna, Puławy
  - Poradnia Kardiologiczna SPZOZ Pulawy, Puławy
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Strawczyński, Płock
  - Indywidualna Specjalistyczna Praktyka Lekarska Magdalena Poterala, Radom
  - Poradnia Kardioogiczna Zegara Słonecznego, Radom
  - Specjalistyczna Praktyka Lekarska Radzionków, Radzionków
  - Indywidualna Specjalistyczna Praktyka Lekarska dr n. med. Alicja Gałuszka-Bilińska, Rybnik
  - Specjalistyczna Praktyka Lekarska Wiesława Faberska-Blicharska, Rybnik
  - Centrum Medyczne Sabamed, Rzeszów
  - Prywatny Gabinet Kardiologiczny dr n.med Janusz Romanek, Rzeszów
  - My Life Centrum chorób serca, Sanok
  - Monika Kujawiak Prywatna Praktyka Lekarska, Siedlce
  - Prywatny Gabinet Lekarski Hanna Wilk-Manowiec, Siedlce
  - Indywidualna praktyka lekarska Artur Marcinkiewicz, Siemianowice Śląskie
  - Asnyka 78d Gabinety Lekarskie, Skierniewice
  - Specjalistyczna Praktyka Lekarska Maciej Kaźmierski, Sosnowiec
  - Specjalistyczna Praktyka Lekarska Marek Kondys, Sosnowiec
  - Powiatowy Szpital Specjalistyczny w Stalowej Woli, Stalowa Wola
  - Centrum Medyczne VITA, Szczecin
  - Specjalistyczna Praktyka Lekarska Tomasz Urbanik, Szczecin
  - ISPL Anna Bis, Szczecin
  - Szpital w Szczecinku, Szczecinek
  - Gabinet Lekarski Weronika Greberska, Szczytniki
  - Specjalistyczna Praktyka Lekarska Kamila Stembalska, Ścinawa
  - Leomed Centrum Medyczne, Tarnowskie Góry
  - Specjalistyczna Praktyka Lekarska Paweł Kocik, Tarnów
  - Prywatna Praktyka Lekarska na wezwanie Mirosław Marciniak, Torun
  - Indywidualna Specjalistyczna Praktyka Lekarska - Witold Orszulak, Tychy
  - Urszula Urbanowicz Specjalistyczna Praktyka Lekarska, Tychy
  - SERCE S.C. Przychodnia Lekarzy Specjalistów, Warsaw
  - Klinika 37 Centrum Kardiologii Płowiecka, Warsaw
  - Prywatny Gabinet Lekarski Bożena Norwa-Otto, Warsaw
  - Gabinet Lekarski lek med. Robert Włodarczyk, Wawrzeńczyce
  - Centrum Medyczne Nowe Miasto, Wałbrzych
  - Specjalistyczny Gabinet Lekarski Łukasz Graczykowski, Włocławek
  - Specjalistyczna Prajtyka Lekarska Grażyna Glanowska, Zabrze
  - Gabinet Prywatnej Praktyki Lekarskiej Kard.-Int . Dr n.med. Brygida Przywara-Chowaniec, Zabrze
  - Ns Zoz Kardiologia Sp. Z.O.O., Zamość
  - ALDEMED Centrum Medyczne, Zielona Góra
  - Gabinety Lekarskie JM Kulczyccy, Żary
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów
  - Poradnia Kardiologiczna Centrum Medyczne w Łańcucie, Łańcut
  - SP ZOZ Łęczna, Łęczna
  - Kardiologiczno - Internistyczny Gabinet Lekarski Skrzyński Andrzej, Łuków
- Romania (106):
  - Miclea Ioana - Mariana MEDIC SPECIALIST CARDIOLOG, Alba Iulia
  - Dr. Morar Mihnea-Dragoscabinet Medical Individual - Specialist Cardiologie, Arad
  - Dr. Pop-Moldovan Adina-Ligia - Medicina Interna - Cardiologie, Arad
  - CMI Iosipescu Laura Cristina, Bacau
  - Cardio Animus SRL, Bacau
  - CMI - Centrul medical Diacord, Baia Mare
  - Mercea Corina-Delia - Medic, Baia Mare
  - Ambrinomed SRL, Botoșani
  - Cardioland SRL, Brasov
  - Rus V. Horatiu - Cabinet Medical Individual de Cardiologie, Brasov
  - S.C. Ilro Medical S.R.L, Bucharest
  - PFA Balahura Cristian, Bucharest
  - Dr. Danet Ruxandra - Medic Cardiologie, Bucharest
  - Dr. Bogdan Stefan Nicolae, Bucharest
  - Cardiocare Center SRL, Bucharest
  - Cordmedica SRL, Bucharest
  - Dr. Serban Irina-Ruxandra - MEDIC PRIMAR CARDIOLOGIE, Bucharest
  - Urocard Plus Srl, Bucharest
  - Medi Pro Consult SRL, Bucharest
  - Cmi Dr Georgescu Dragos, Bucharest
  - Dr. Geavlete Dana-Oliviana - Activitate Medicala, Bucharest
  - Mihaila I. Sorina - Medic Pfi, Bucharest
  - S.C. Cardiomedical Team Pro S.R.L., Bucharest
  - Dumitrescu Silviu-Ionel Persoana Fizica Autorizata, Bucharest
  - Mihalcea Janina-Diana Medic Specialist Cardiologie, Bucharest
  - Patrascu R. Natalia - Medic Specialist Medicina Interna, Bucharest
  - Popescu I. Ileana Nicoleta Medic specialist cardiologie, Bucharest
  - CMI Dr. Parsa Motlagh Babak, Bucharest
  - Magister Research SRL, Bucharest
  - Dr. Lungeanu-Juravle Laura-Activitate Medicala, Bucharest
  - Cardio Clinique NCS SRL, Buzău
  - Medcon SRL, Buzău
  - Medicard SRL, Buzău
  - Angioplast Medical srl, Ciurea
  - CMI Diaconescu Iulia Dana, Cluj-Napoca
  - Mediprax Centrum Cluj Napoca, Cluj-Napoca
  - SC Adisan SRL, Cluj-Napoca
  - Sc Medicardio Andreea Srl, Cluj-Napoca
  - Cardiotreat SRL, Cluj-Napoca
  - SC Clujana Medica Srl, Cluj-Napoca
  - PFA Comsa M.Dan-Horatiu, Cluj-Napoca
  - Cabinet Cardiohealt Srl, Cluj-Napoca
  - SC Cardioprotect MED SRL, Cluj-Napoca
  - Sc Dentcor Srl, Cluj-Napoca
  - Cardio World Health, Com Mosoaia
  - Cardio Manea Adelina SRL, Constanța
  - Endodiahealth Srl, Constanța
  - Dr. Maxim George Razvan - Activitate Medicala, Constanța
  - CMI Dr Ilie Ivona Valeria, Constanța
  - Asclepios Medicalhealth SRL, Constanța
  - Sc Daxiela Impex Srl, Craiova
  - Hortopan Med SRL, Craiova
  - Neurocord Medical Srl, Craiova
  - Vesalius Medical S.R.L, Craiova
  - Cabinet Medical Individual - Dr. Popescu Monica, Craiova
  - SC A&C Medical Prime SRL, Craiova
  - S & R Cardiobalance Srl, Curtea de Argeş
  - Cardiolife, Deva
  - Bendl H. Laura Elena - Cabinet Medical Individual Plus Clinic, Drobeta-Turnu Severin
  - SC Maycor SRL, Galati
  - CMI Dr. Chiscaneanu Teodor, Galati
  - Cardiomedplus SRL, Gheorghieni
  - Procardia Serv-Med 2009 SRL srl, Iași
  - Sc Cardiocare Clinic Srl, Iași
  - Sc Cardiortomed Srl, Iași
  - Medical Cardio Anghel SRL, Iași
  - Niculescu G. Ana Irina - Medic colaborator, Iași
  - SC Cardiomed SRL Iasi, Iași
  - Cardioszakacs Srl, Cui 34404518, Miercurea-Ciuc
  - Polimed Center SRL, CUI 26072639, Odorheiu Secuiesc
  - CMI Dr. Rotariu Dragos, Oradea
  - CMI Societatea civila Magheru&Magheru, Oradea
  - CMI Cardiomed SRL, Oradea
  - PFA Dr. Ardelean Adriana Ioana, Oradea
  - Dradiand SRL, Oradea
  - Sc Adriacard Srl, Oradea
  - Simed Concept SRL, Ostratu
  - Andries I. Elena - Medic Primar Cardiologie Si Medic Specialist Mi, Piatra Neamţ
  - Cardiomed Alexandrescu Srl-D, Piatra Neamţ
  - Dr. Corcoz Cardiologie SRL, Piatra Neamţ
  - Davisof San Srl, Piteşti
  - Clinica Cardiologie Dr Stanciu Viorel, Piteşti
  - Sc Procordia Concept Srl, Piteşti
  - Cavi Clinique SRL, Ploieşti
  - SC Cardiologie Dr. Cristina Radoi SRL, Râmnicu Vâlcea
  - Sc Lidermed Plus Srl, Râmnicu Vâlcea
  - Sc Incarmed Srl, Râmnicu Vâlcea
  - Munteanu Alice-Elena - Medic Cardiolog, Sat Rosu, Comuna Chiajna
  - Cardio Stim Center SRL, Sânpetru
  - Gx.Hatconsulting Srl, Săcele
  - Voineag Olivia Medic Colaborator, Scheia
  - SC Endocordis SRL, Sfântu Gheorghe
  - Rusu N. Ramona Iulia Medic Primar Cardiologie, Suceava
  - Batar D. Sergiu Constantin, Şelimbăr
  - German Sallo Marta - Medic primar cardiolog, CIF 35699735, Târgu Mureş
  - CMI Tatar A. Maria Cristina, CUI 19814204, Târgu Mureş
  - Diaconu Diana - Medic Cif 31885867, Tifgu Mures
  - Cardiomed Health SRL, Timișoara
  - Mornos Cristian Medic Independent, Timișoara
  - Cardio Suport SRL, Timișoara
  - Medicalife Tim SRL, Timișoara
  - Cardio - DRS S.R.L, Timișoara
  - Policlinica Dr. Tudoran, Timișoara
  - Croitoru G Rodica Medic Colaborator, Valea Adâncă
  - CMI Demle S. Adriana-Cristina, Zalău
  - Dr. Dragos Lupu - Medic Specialist Cardiolog, Zarnesti
- Switzerland (39):
  - Universitätsspital Basel, Basel
  - Spital Sonnenhof, Bern
  - Engeried-Spital (Bern), Bern
  - Spitalzentrum Biel, Biel
  - Hôpital de La Tour, Carouge
  - Cardiomed - Jura, Courrendlin
  - Centre de Cardiologie, Delémont
  - Schlossberg Ärztezentrum, Frauenfeld
  - Hôpitaux Universitaires de Genève, Geneva
  - Spital Lachen AG, Lachen
  - CHUV-Centre hospitalier universitaire vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Herzzentrum Hirslanden Zentralschweiz, Lucerne
  - Hôpital de Morges, Morges
  - Dr. med. Eleni Goulouti, Neuchâtel
  - Kantonsspital Olten, Olten
  - Herzpraxis Regensdorf, Regensdorf
  - Herzpraxis Sankt Gallen, Sankt Gallen
  - Kantonsspital Obwalden, Sarnen
  - Rehaklinik Seewis, Seewis
  - Dr. med. Kiril Tzvetanov, Sierre
  - Herzpraxis Sursee, Sursee
  - Kardiologie Aarezentrum Thun, Thun
  - Spital STS AG, Thun
  - Hôpital Fribourgeois, Villars-sur-Glâne
  - Herz- und Physiozentrum, Wallisellen
  - Arztpraxis Waltenschwil, Waltenschwil
  - Spital Will, Will
  - Herz- und Kreislaufpraxis Winterthur, Winterthur
  - Medbase Winterthur Neuwiesen, Winterthur
  - Hôpital d'Yverdon-les-Bains, Yverdon-les-Bains
  - Spital Zollikerberg, Zollikerberg
  - SICADE Clinic, Zurich
  - Herzpraxis Enge ZH, Zurich
  - Gruppenpraxis Dr. Deseö / Dr. Deseö-Schütz / Dr. Lorger, Zurich
  - Herzklinik Hirslanden, Zurich
  - HerzKlinik Zürich Hirslanden, Zurich
  - Herzkreislaufpraxis, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multinational, non-interventional study based on newly collected data to assess the demographics and treatment patterns of patients with heart failure (HF), with or without diabetes, using a two-cohort design: one cohort included patients with a first prescription of empagliflozin as routine therapy for HF, while the other cohort included patients receiving drugs with a mechanism of action different from empagliflozin.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a group if any of the entry criteria were violated.
Period: Visit 1 - Baseline
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients
Started (Patients recruited) | 3327 | 104
Full Analysis Set (FAS) | 3320 | 104
Treated (Receiving a drug prescription) | 3309 | 104
Completed | 3309 | 104
Not Completed | 18 | 0
Not completed — Not-treated | 18 | 0
Period: Visit 1 to Visit 2 - 24 Weeks
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients
Started | 3309 | 0 (Non-SGLT2i-treated patients were not followed past Visit 1.)
Completed | 3152 | 0
Not Completed | 157 | 0
Not completed — Still active/screening failure | 25 | 0
Not completed — Other reason than listed | 36 | 0
Not completed — Death | 45 | 0
Not completed — Adverse-drug reaction/heart failure hospitalization | 7 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 38 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: all registered patients who gave informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients | Total
Number analyzed (Participants) | 3320 | 104 | 3424
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.63 (10.52) | 79.67 (10.56) | 69.67 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1224 | 47 | 1271
  Male | 2096 | 57 | 2153
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: Units on a scale] — The KCCQ includes 23 items across 7 domains: physical limitation, symptom stability, symptom frequency and burden, self-efficacy, quality of life, and social limitation. The total symptom score (TTS) is calculated as the mean of the symptom-related scores. The clinical summary score (CSS) is calculated as the mean of the physical limitation and total symptom score. The overall symptom score (OSS) is calculated as the mean of the physical limitation, total symptom, quality of life, and social limitation score. All scores range from 0 to 100, with higher scores indicating better health. Population: Full analysis set: all registered patients who gave informed consent. Patients without baseline KCCQ values were excluded.
  Units on a scale
    CSS: number analyzed (Participants) | 3314 | 103 | 3417
    CSS | 61.64 (22.45) | 67.23 (17.90) | 61.81 (22.35)
    TSS: number analyzed (Participants) | 3314 | 103 | 3417
    TSS | 59.03 (24.86) | 66.13 (20.57) | 59.25 (24.76)
    OSS: number analyzed (Participants) | 3314 | 103 | 3417
    OSS | 56.29 (22.73) | 61.46 (20.21) | 56.45 (22.67)

OUTCOME MEASURES:

1. Primary Outcome: Change of the Kansas City Cardiomyopathy Questionnaire (KCCQ) Scores in Patients Newly Treated With Empagliflozin According to Routine Practice
Description: Change from baseline to Week 24 of the Kansas City Cardiomyopathy Questionnaire (KCCQ) scores, calculated as [Week 24] - [Baseline]. The KCCQ includes 23 items across 7 domains: physical limitation, symptom stability, symptom frequency, symptom burden, self-efficacy, quality of life, and social limitation. This outcome measured the total symptom score (TTS), clinical summary score (CSS), and overall summary score (OSS) in the empagliflozin-treated patients as defined in the clinical study protocol. The TTS evaluates symptom frequency and burden and is calculated as the mean of the symptom frequency score and symptom burden score. The CSS is calculated as the mean of the physical limitation score and total symptom score. The OSS is calculated as the mean of the physical limitation score, total symptom score, quality of life score, and social limitation score. The TTS, CSS, and OSS are represented on a 0-to-100-point scale, where a higher score reflects better health status.
Time Frame: At baseline and at week 24.
Population: Primary endpoint set (PES): All patients, who received at least one dose of empagliflozin for HF and have filled in KCCQ at baseline and week 24.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Empagliflozin-treated Patients
Number analyzed (Participants) | 3108
Units on a scale
  CSS | 14.66 (18.44)
  TSS | 17.61 (21.04)
  OSS | 16.47 (18.86)

2. Secondary Outcome: Change of the New York Heart Association (NYHA) Class in Patients Newly Treated With Empagliflozin
Description: This outcome measured the number of patients newly treated with empagliflozin who experienced a change in the New York Heart Association (NYHA) Class from baseline to Week 24. The NYHA Classes of heart failure categorize patients with symptomatic or advanced heart failure based on their physical activity limitations. Class I patients present no limitation of physical activity, and ordinary physical activity does not cause fatigue, palpitations, or shortness of breath. Class II patients present a slight limitation of physical activity, characterized by fatigue, palpitations, shortness of breath, or chest pain as a result of ordinary physical activity. Class III patients are characterized by a marked limitation of physical activity, where less than ordinary activity causes fatigue, palpitations, shortness of breath, or chest pain. Class IV patients present symptoms of heart failure at rest, where any physical activity causes further discomfort.
Time Frame: At baseline and at Week 24.
Population: Safety set (SAF): All patients of FAS who received empagliflozin at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin-treated Patients
Number analyzed (Participants) | 3309
Participants
  Baseline Class II: number analyzed (Participants) | 1981
  Baseline Class II: Week 24 Class I | 337
  Baseline Class II: Week 24 Class II | 1388
  Baseline Class II: Week 24 Class III | 54
  Baseline Class II: Week 24 Class IV | 0
  Baseline Class II: Unknown | 5
  Baseline Class II: Missing | 184
  Baseline Class II: No Week 24 visit | 13
  Baseline Class III: number analyzed (Participants) | 1263
  Baseline Class III: Week 24 Class I | 37
  Baseline Class III: Week 24 Class II | 730
  Baseline Class III: Week 24 Class III | 368
  Baseline Class III: Week 24 Class IV | 3
  Baseline Class III: Unknown | 0
  Baseline Class III: Missing | 118
  Baseline Class III: No Week 24 visit | 7
  Baseline Class IV: number analyzed (Participants) | 64
  Baseline Class IV: Week 24 Class I | 0
  Baseline Class IV: Week 24 Class II | 20
  Baseline Class IV: Week 24 Class III | 22
  Baseline Class IV: Week 24 Class IV | 10
  Baseline Class IV: Unknown | 0
  Baseline Class IV: Missing | 12
  Baseline Class IV: No Week 24 visit | 0
  Baseline Missing: number analyzed (Participants) | 1
  Baseline Missing: Week 24 Class I | 0
  Baseline Missing: Week 24 Class II | 0
  Baseline Missing: Week 24 Class III | 0
  Baseline Missing: Week 24 Class IV | 0
  Baseline Missing: Unknown | 0
  Baseline Missing: Missing | 1
  Baseline Missing: No Week 24 visit | 0

3. Secondary Outcome: Number of Participants With Comorbidities
Description: Number of patients with first prescription of empagliflozin and patients prescribed drugs other than SGLT2 inhibitors with concomitant disease/comorbidities. Concomitant diseases/comorbidities are presented according to the ICD-10-CM (the International Classification of Diseases, Tenth Revision, Clinical Modification) standardized system using the disease code.
Time Frame: At baseline.
Population: FAS: All registered patients who gave informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients
Number analyzed (Participants) | 3320 | 104
Participants
  E03.- Other hypothyroidism | 130 | 6
  E10.- Insulin-dependent diabetes mellitus | 103 | 3
  E11.- Non-insulin-dependent diabetes mellitus | 626 | 18
  E66.- Obesity | 265 | 6
  E78.- Disorders of lipoprotein metabolism and other lipidaemias | 1197 | 49
  E79.- Disorders of purine and pyrimidine metabolism | 188 | 3
  I10 Essential (primary) hypertension | 1380 | 54
  I11.- Hypertensive heart disease | 604 | 21
  I20.- Angina pectoris | 291 | 8
  I21.- Acute myocardial infarction | 186 | 3
  I25.- Chronic ischaemic heart disease | 1164 | 25
  I27.- Other pulmonary heart diseases | 56 | 4
  I34.- Nonrheumatic mitral valve disorders | 517 | 30
  I35.- Nonrheumatic aortic valve disorders | 215 | 18
  I36.- Nonrheumatic tricuspid valve disorders | 174 | 11
  I42.- Cardiomyopathy | 256 | 8
  I44.- Atrioventricular and left bundle-branch block | 139 | 5
  I48 Atrial fibrillation and flutter | 1183 | 27
  I49.- Other cardiac arrhythmias | 132 | 4
  I70.- Atherosclerosis | 116 | 2
  J44.- Other chronic obstructive pulmonary disease | 117 | 4
  N18.- Chronic kidney disease | 211 | 6
  N40 Hyperplasia of prostate | 119 | 1
  Z95.- Presence of cardiac and vascular implants and grafts | 547 | 15

4. Secondary Outcome: Number of Participants With Concomitant Heart-failure (HF) Related Medication
Description: Number of patients who took concomitant HF-related medication.
Time Frame: At baseline.
Population: FAS: All registered patients who gave informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients
Number analyzed (Participants) | 3320 | 104
Participants
  Acetylsalicylic acid | 63 | 4
  Bisoprolol | 868 | 19
  Candesartan | 68 | 4
  Carvedilol | 233 | 2
  Eplerenone | 517 | 5
  Furosemide | 913 | 31
  Indapamide | 58 | 5
  Metoprolol | 457 | 11
  Nebivolol | 98 | 6
  Perindopril | 207 | 9
  Ramipril | 413 | 6
  Sacubitril | 112 | 0
  Sacubitril and valsartan | 443 | 5
  Spironolactone | 981 | 20
  Torasemide | 645 | 5
  Valsartan | 166 | 0

5. Secondary Outcome: Hospitalizations Due to Heart-failure in the Past 6 Months Before Baseline
Description: Number of patients hospitalized at least one time due to heart failure (HF).
Time Frame: Up to 6 months prior to baseline visit.
Population: FAS: All registered patients who gave informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin-treated Patients | Non-SGLT2i-treated Patients
Number analyzed (Participants) | 3320 | 104
Participants | 284 | 6

ADVERSE EVENTS:
Time Frame: From start of empagliflozin to its last administration plus 7 days. Up to 25 weeks.
Description: Safety set: All registered patients who gave informed consent and who received empagliflozin at least once.
  As per protocol, patients not receiving empagliflozin were not observed past Visit 1, and adverse events were not collected.
Arm/Group | Empagliflozin-treated Patients
All-Cause Mortality (participants affected / at risk) | 46/3309
Serious Adverse Events (participants affected / at risk) | 74/3309
Other Adverse Events (participants affected / at risk) | 0/3309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin-treated Patients (N=3309)
Death (General disorders) | 17
Cardiac failure (Cardiac disorders) | 14
Cardiac arrest (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 3
Sudden cardiac death (General disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Hospitalisation (Surgical and medical procedures) | 2
Myocardial infarction (Cardiac disorders) | 2
Sudden death (General disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Blood pressure increased (Investigations) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Escherichia pyelonephritis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Necrotising fasciitis (Infections and infestations) | 1
Necrotising oesophagitis (Gastrointestinal disorders) | 1
Performance status decreased (General disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Polyneuropathy (Nervous system disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT05350202/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT05350202/SAP_001.pdf